CLINICAL TRIAL: NCT02521493
Title: Risk-Stratified Therapy for Acute Myeloid Leukemia in Down Syndrome
Brief Title: Response-Based Chemotherapy in Treating Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndrome in Younger Patients With Down Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAML1531; NCI-2015-00324 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML1531; s16-01673; AAML1531 (Other: Children's Oncology Group); AAML1531 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Results first posted 2025-06-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Down Syndrome; Myelodysplastic Syndrome; Myeloid Leukemia Associated With Down Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Down Syndrome; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Asparaginase; Leyk; asparaginase erwinia chrysanthemi recombinant; Cytarabine; Daunorubicin; Etoposide; Mitoxantrone; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (standard risk) (Experimental): INDUCTION II: Patients receive cytarabine IV continuously over 96 hours, daunorubicin hydrochloride IV over 1-15 minutes, and thioguanine PO BID on days 1-4. Induction II continues for a minimum of 28 days.
  INDUCTION III: Patients receive cytarabine, daunorubicin hydrochloride, and thioguanine as in Induction II. Induction III continues for a minimum of 28 days.
  INTENSIFICATION I: Patients receive cytarabine IV continuously over 168 hours on days 1-7 and etoposide IV over 60-120 minutes on days 1-3. Intensification I continues for a minimum of 28 days.
  INTENSIFICATION II: Patients receive cytarabine and etoposide as in Intensification I. Intensification II continues for a minimum of 28 days.
  (This arm is closed to accrual and treatment with amendment #4A 01/07/2019)
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Thioguanine
- Arm B (high risk) (Experimental): INDUCTION II: Patients receive high dose cytarabine IV over 1-3 hours Q12 hours on days 1-4 and mitoxantrone hydrochloride IV over 15-30 minutes on days 3-6. Induction II continues for a minimum of 28 days.
  INTENSIFICATION I: Patients receive high dose cytarabine IV over 1-3 hours Q12 hours and etoposide IV over 90-120 minutes on days 1-5. Intensification I continues for a minimum of 28 days.
  INTENSIFICATION II: Patients receive high dose cytarabine IV over 3 hours Q12 hours on days 1, 2, 8, and 9. Patients also receive asparaginase or asparaginase Erwinia chrysanthemi IM or IV over 30 minutes on days 2 and 9. Intensification II continues for a minimum of 28 days.
  Interventions: Drug: Asparaginase; Drug: Asparaginase Erwinia chrysanthemi; Drug: Cytarabine; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: Asparaginase — Given IM or IV
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-Asparaginase; L-Asparagine Amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa; Spectrila
  Arms: Arm B (high risk)
Drug: Asparaginase Erwinia chrysanthemi — Given IM or IV
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
  Arms: Arm B (high risk)
Drug: Cytarabine — Given IT and IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: Arm A (standard risk)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: Arm A (standard risk)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
  Arms: Arm B (high risk)
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Arm A (standard risk)

SUMMARY:
This phase III trial studies response-based chemotherapy in treating newly diagnosed acute myeloid leukemia or myelodysplastic syndrome in younger patients with Down syndrome. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Response-based chemotherapy separates patients into different risk groups and treats them according to how they respond to the first course of treatment (Induction I). Response-based treatment may be effective in treating acute myeloid leukemia or myelodysplastic syndrome in younger patients with Down syndrome while reducing the side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 2-year event-free-survival (EFS) for children with standard risk Down syndrome (DS) acute myeloid leukemia (AML) (minimal residual disease [MRD]-negative after one cycle of induction therapy) after elimination of high dose (HD) Ara-C (cytarabine) from the treatment regimen.

II. To determine the 2-year EFS for children with high risk DS AML (MRD-positive after one cycle of induction therapy) after intensification of treatment equivalent to that used for high risk AML in children without DS.

EXPLORATORY OBJECTIVES:

I. To compare the feasibility and analytical characteristics of flow cytometry, polymerase chain reaction (PCR) and targeted error-corrected sequencing of GATA binding protein 1 (globin transcription factor 1) (GATA1) mutations as methods to detect MRD in DS AML.

II. To establish a DS AML cell bank of viably frozen bone marrow samples collected at the end of induction and corresponding non-tumor deoxyribonucleic acid (DNA) samples collected at end of Induction 1.

OUTLINE:

INDUCTION I: Patients receive cytarabine intrathecally (IT) on day 1 and intravenously (IV) continuously over 96 hours, daunorubicin hydrochloride IV over 1-15 minutes, and thioguanine orally (PO) twice daily (BID) on days 1-4. Induction I continues for a minimum of 28 days.

Patients are assigned to 1 of 2 treatment arms based on their MRD status after completion of Induction I.

ARM A (STANDARD RISK) (Closed to accrual and treatment with amendment #4A 01/07/2019):

INDUCTION II: Patients receive cytarabine IV continuously over 96 hours, daunorubicin hydrochloride IV over 1-15 minutes, and thioguanine PO BID on days 1-4. Induction II continues for a minimum of 28 days.

INDUCTION III: Patients receive cytarabine, daunorubicin hydrochloride, and thioguanine as in Induction II. Induction III continues for a minimum of 28 days.

INTENSIFICATION I: Patients receive cytarabine IV continuously over 168 hours on days 1-7 and etoposide IV over 60-120 minutes on days 1-3. Intensification I continues for a minimum of 28 days.

INTENSIFICATION II: Patients receive cytarabine and etoposide as in Intensification I. Intensification II continues for a minimum of 28 days.

ARM B (HIGH RISK):

INDUCTION II: Patients receive high dose cytarabine IV over 1-3 hours every 12 (Q12) hours on days 1-4 and mitoxantrone hydrochloride IV over 15-30 minutes on days 3-6. Induction II continues for a minimum of 28 days.

INTENSIFICATION I: Patients receive high dose cytarabine IV over 1-3 hours Q12 hours and etoposide IV over 90-120 minutes on days 1-5. Intensification I continues for a minimum of 28 days.

INTENSIFICATION II: Patients receive high dose cytarabine IV over 3 hours Q12 hours on days 1, 2, 8, and 9. Patients also receive asparaginase or asparaginase Erwinia chrysanthemi (E. carotovora) intramuscularly (IM) or IV over 30 minutes on days 2 and 9. Intensification II continues for a minimum of 28 days.

After completion of study treatment, patients are followed up at 1 month, monthly for 12 months, every 3 months for 12 months, every 6 months for 3 years, annually for 10 years, and in case of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have constitutional trisomy 21 (Down syndrome) or trisomy 21 mosaicism (by karyotype or fluorescence in situ hybridization [FISH])
* Patient has one of the following:

  * Patient has previously untreated de novo AML and meets the criteria for AML with >= 20% bone marrow blasts as set out in the World Health Organization (WHO) Myeloid Neoplasm classification

    * Attempts to obtain bone marrow either by aspirate or biopsy must be made unless clinically prohibitive; in cases where it is clinically prohibitive, peripheral blood with an excess of 20% blasts and in which adequate flow cytometric and cytogenetics/FISH testing is feasible can be substituted for the marrow exam at diagnosis
  * Patient has cytopenias and/or bone marrow blasts but does not meet the criteria for the diagnosis of AML (WHO Myeloid Neoplasm classification) because of < 20% marrow blasts and meets the criteria for a diagnosis of myelodysplastic syndrome (MDS)
  * For patients who do not meet criteria for AML or MDS as outlined above; patient has a history of transient myeloproliferative disorder (which may or may not have required chemotherapy intervention and:

    * Is > 8 weeks since resolution of transient myeloproliferative disease (TMD) with >= 5% blasts, OR
    * Has an increasing blast count (>= 5%) in serial bone marrow aspirates performed at least 4 weeks apart
* Children who have previously received chemotherapy, radiation therapy or any anti-leukemic therapy are not eligible for this protocol, with the exception of cytarabine for the treatment of TMD
* There are no minimal organ function requirements for enrollment on this study

  * Note: Previous cardiac repair with sufficient cardiac function is not an exclusion criteria
* Each patient's parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human subjects research must be met

Exclusion Criteria:

* Patients with promyelocytic leukemia (French-American-British [FAB] M3)
* Prior therapy

  * Patients =< 30 days from the last dose of cytarabine used for treatment of TMD

Ages: 91 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jason N Berman, Principal Investigator — Children's Oncology Group
Locations (191):
- United States (169):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (11):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Berman JN, Verma A, Viola SA, Alonzo T, Wang YC, Brodersen LE, Loken MR, Beckman AK, Hirsch BA, Raimondi S, Chisholm KM, Ma X, Ries RE, Meshinchi S, Gamis AS, Schore RJ, Taub JW, Kolb EA, Cooper TM, Hitzler JK. Molecular Risk Markers Define Risk of Relapse in Myeloid Leukemia of Down syndrome Beyond Measurable Residual Disease. Blood Adv. 2025 Oct 22:bloodadvances.2025017837. doi: 10.1182/bloodadvances.2025017837. Online ahead of print. PMID 41124669
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Standard Risk): Patients with MRD <0.05%
  (This arm was closed to accrual and treatment with amendment #4A 01/07/2019)
- Arm B (High Risk): Patients with MRD ≥ 0.05%
- No Risk Stratification: No Risk Stratification
Period: Overall Study
Arm/Group | Arm A (Standard Risk) | Arm B (High Risk) | No Risk Stratification
Started | 114 | 44 | 122
Completed | 89 | 38 | 0
Not Completed | 25 | 6 | 122
Not completed — Death | 3 | 4 | 1
Not completed — Physician Decision | 19 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0
Not completed — Post Amd4A (MRD < 0.05%) | 0 | 0 | 115
Not completed — No MRD result | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Standard Risk) | Arm B (High Risk) | No Risk Stratification | Total
Number analyzed (Participants) | 114 | 44 | 122 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 114 | 44 | 122 | 280
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.7 (0.7) | 1.7 (0.6) | 1.7 (0.8) | 1.7 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 21 | 61 | 142
  Male | 54 | 23 | 61 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 3 | 33 | 66
  Not Hispanic or Latino | 78 | 33 | 82 | 193
  Unknown or Not Reported | 6 | 8 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 5 | 3 | 10 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 16 | 9 | 19 | 44
  White | 72 | 24 | 70 | 166
  More than one race | 3 | 0 | 2 | 5
  Unknown or Not Reported | 16 | 8 | 19 | 43
Region of Enrollment [Number; unit: participants]
  United States | 108 | 38 | 108 | 254
  Canada | 3 | 5 | 7 | 15
  Australia | 1 | 1 | 5 | 7
  New Zealand | 2 | 0 | 1 | 3
  Saudi Arabia | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: The Kaplan-Meier method will be used to estimate 2-year EFS separately for standard risk and high risk patients. EFS is defined as the time from the end of Induction I to failure to achieve remission at the end of Induction II, relapse, occurrence of a second malignancy, or death.
Time Frame: Up to 2 years from study entry
Population: The High Risk Arm excludes the following patients: 1 Ineligible, 1 withdrawal, 1 death prior to Induction II. The No Risk Stratification Arm had zero patients for induction II treatment, as all patients went off study at the end of Induction I
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Standard Risk) | Arm B (High Risk)
Number analyzed (Participants) | 114 | 41
percentage of patients | 89.37 [82 to 93.8] | 80.49 [64.8 to 89.7]

2. Other Pre Specified Outcome: Mean Length on Protocol Therapy
Description: The mean number of days patients spent on protocol therapy.
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Proportion of Patients With an Early Death
Description: The proportion of patients experiencing an early death in the first month.
Time Frame: Up to 1 month from study entry
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate 2-year OS defined as the time from the end of Induction I to death.
Time Frame: Up to 2 years from study entry
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Proportion With Treatment Related Mortality
Description: The proportion of patients experiencing a treatment related death will be reported along with a corresponding confidence interval.
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Proportion of Patients Experiencing a Relapse Risk
Description: The proportion of patients experiencing a relapse after achieving remission will be reported along with a corresponding confidence interval.
Time Frame: Up to 2 years from study entry
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Percentage of Patients Experiencing Grade 3+ Adverse Events (AE)
Description: The percentage of patients experiencing grade 3 or higher AEs will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Mean Time to Absolute Neutrophil Count (ANC) Recovery
Description: The mean time to recovery of ANC to at least 1000/uL will be reported.
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Mean Duration of Hospitalization
Description: Mean number of days patients are hospitalized.
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Proportion of Patients With at Least 1 Infection
Description: The proportion of patients having at least one infection will be reported.
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: While patients were on Protocol Therapy: Up to 5 courses, 28-day cycles
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Arm A (Standard Risk) | Arm B (High Risk) | No Risk Stratification
All-Cause Mortality (participants affected / at risk) | 12/114 | 8/43 | 1/122
Serious Adverse Events (participants affected / at risk) | 3/114 | 1/43 | 2/122
Other Adverse Events (participants affected / at risk) | 84/114 | 37/43 | 54/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Standard Risk) (N=114) | Arm B (High Risk) (N=43) | No Risk Stratification (N=122)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Infections and infestations - Other, specify: Metapneumovirus (Infections and infestations) | 0 | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Standard Risk) (N=114) | Arm B (High Risk) (N=43) | No Risk Stratification (N=122)
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 12 | 7 | 8
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 2 | 0 | 0
Anal pain (Gastrointestinal disorders) | 0 | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 13 | 5 | 2
Anorexia (Metabolism and nutrition disorders) | 9 | 8 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 6 | 4
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 1
Catheter related infection (Infections and infestations) | 6 | 4 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 20 | 3 | 4
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 5 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 39 | 22 | 27
Fever (General disorders) | 2 | 5 | 1
Fibrinogen decreased (Investigations) | 0 | 0 | 1
GGT increased (Investigations) | 2 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 3 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 4 | 4 | 3
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 6 | 8 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypotension (Vascular disorders) | 2 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 3
Infections and infestations - Other, specify (Infections and infestations) | 22 | 11 | 4
Infusion site extravasation (General disorders) | 1 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 2 | 6 | 0
Lymphocyte count decreased (Investigations) | 3 | 4 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 5 | 7
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 17 | 7 | 2
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 17 | 5 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary valve disease (Cardiac disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 6 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 5 | 7
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin infection (Infections and infestations) | 3 | 3 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Small intestine infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Stoma site infection (Infections and infestations) | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 5 | 6 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0
Vulval infection (Infections and infestations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 11 | 6 | 1
Wound infection (Infections and infestations) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02521493/Prot_SAP_000.pdf